CLINICAL TRIAL: NCT01428804
Title: Pilot Study of Feasibility of the Effect of Treatment With tDCS in Patients Suffering From Resistant Depression
Brief Title: Study of Transcranial Direct Current Stimulation (tDCS) as add-on Treatment for Resistant Major Depression
Acronym: DEPRESCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEPRESCO
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Resistant Major Depression
Keywords: Resistant Major Depression; Mood disorders; tDCS
MeSH Terms: conditions — Mood Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Active Comparator): a group named G1 and treated by medication with escitalopram (Seroplex®) stabilized for at least 1 month and 10 sessions of tDCS anode active at 2 sessions per day (1 morning and 1 afternoon) for 5 days with an electric current 2 mA
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- sham tDCS (Sham Comparator): a group named G2 and treated by medication with escitalopram (Seroplex®) stabilized for at least 1 month and sham tDCS.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — Device: Eldith DC-Stimulator real or sham tDCS for 20 minutes at 2mA intensity over the left DLPFC (F3 according to the 10-20 system) Other Name: Eldith DC - Stimulator (neuroConn GmbH, Ilmenau, Germany)
  Other Names: Eldith DC - Stimulator (neuroConn GmbH, Ilmenau, Germany)

SUMMARY:
The purpose of the study is to investigate the effect of tDCS applied at the anodic left DLPFC of patients with resistant depression compared to patients treated with conventional therapy. The tDCS is used in add-on drug treatment with antidepressants of reference in resistant depression.

DETAILED DESCRIPTION:
The aim of our study is to investigate the effect of tDCS applied at the anodic left dorsolateral prefrontal cortex (DLPFC)of patients with resistant depression compared to patients treated with conventional therapy. The tDCS is used in add-on drug treatment with antidepressants of reference in resistant depression.

This is a randomized 2-arm parallel, double blind study comparing 2 groups of 12 patients: patients treated with sham tDCS and whose medication reference is stabilized for a month vs. patients treated by active tDCS 10 sessions over five days and whose medication reference is stabilized for a month. The 24 patients with resistant depression will be selected in the psychiatric department of the University Hospital of Besançon. After giving informed consent, patients will be evaluated by a psychiatrist using the Montgomery Asberg Depression Rating Scale (MADRS), the Hamilton Depression Rating Scale (HDRS), State-Trait Anxiety Inventory (STAI) and Beck Depression Inventory (BDI). The complete assessment takes 40 minutes.

After locating the left DLPFC, treatment with active tDCS with a current of 2 mA or sham will be directed by 20-minute session. A psychometric assessment will be conducted again at the end of treatment week and one month, three months and finally six months after stopping treatment. Scales of comfort and acceptability will also be proposed to the patient to determine whether any gene is caused by this treatment.

This study will include two parallel arms:

* a group named G1 and treated by medication with escitalopram (Seroplex®) stabilized for at least 1 month and 10 sessions of tDCS anode active at 2 sessions per day (1 morning and 1 afternoon) for 5 days with an electric current 2 mA;
* a group named G2 and treated by medication with escitalopram (Seroplex®) stabilized for at least 1 month and sham tDCS.

These two groups are matched for age (+/- 5 years) and gender. The population of this study will be comprised of patients over age 18 with unipolar depressive episode resistant episode characterized by the failure of two antidepressant treatments for depressive episode and treated by medication with escitalopram (Seroplex®) (20 mg/day), since at least 1 month. The delay of one month is a minimum to observe a non-response. Moreover, in term of ethical point of view, it's difficult to wait 6 to 8 weeks to observe the non-response to treatment.

These people will be recruited on a voluntary basis, after notification and consent in the research center, the Psychiatry Clinical Department of the University Hospital of Besançon. This study was conducted over a period of 15 months.

ELIGIBILITY:
Inclusion Criteria:

* subject whose MDD are single or recurrent without psychotic features according to DSM-IV-TR
* subject with a diagnosis of resistant major depression (1 or 2 failed antidepressant treatments for the current depressive episode)
* MADRS score ≥ 25
* subjects with drug treatment by escitalopram (Seroplex®) for at least one month
* right-handed patients
* without severe progressive somatic pathology (especially tumor diseases, degenerative diseases)
* without severe cognitive impairment making psychometric evaluation impossible
* excepted antidepressant treatment, psychotropic following are tolerated during the course of the study : benzodiazepine anxiolytics (up to 20mg/day diazepam equivalent) ; hydroxyzine (up to 50 mg/day) ; cyamemazine (up to 50 mg/day) ; hypnotics (imidazopyridine up to 7.5 mg/day).

Exclusion Criteria:

* subject treated with antipsychotics or mood stabilizers
* subjects resistant to escitalopram (Seroplex®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
MADRS [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk] | [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk]
  The changes in MADRS will constitute the major research outcome measure used to assess response to tDCS

SECONDARY OUTCOMES:
HDRS-21 | [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk]
BDI-13 | [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk]
subscores for anxiety depression scale from HRDS-21 | [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk]
STAI | [time frame: baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk]

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel HAFFEN, Prof., Principal Investigator — CHU Besancon - Clinical Psychiatric Department
Locations (1):
- CHU Besancon - Clinical Psychaitric Department, Besançon, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennabi D, Nicolier M, Monnin J, Tio G, Pazart L, Vandel P, Haffen E. Pilot study of feasibility of the effect of treatment with tDCS in patients suffering from treatment-resistant depression treated with escitalopram. Clin Neurophysiol. 2015 Jun;126(6):1185-1189. doi: 10.1016/j.clinph.2014.09.026. Epub 2014 Oct 5. PMID 25454337